CLINICAL TRIAL: NCT01843907
Title: Cross-sectorial Patient Participation in Prevention of Loss of Functions in Older Short-stay Medical Patients
Brief Title: Patient Participation in Prevention of Loss of Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Tove Lindhardt Damsgaard, Senior Researcher, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-1-2012-118
Record Dates: First submitted 2013-03-20; First posted 2013-05-01 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Dementia; Malnutrition; Depression; Pain; Quality of Life
MeSH Terms: conditions — Dementia; Malnutrition; Depression; Pain | interventions — Nurses

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Empowerment (Other): Patients in the intervention group 1 receive a communication report which will also be sent to the physician and home care. In communication report includes the results and interpretation and explanation of the measurements in layman's terms. The report also includes relevant and targeted information on pain management, depression among the elderly, dementia and disability in old age and ways to maintain and improve functional capacity. Links and addresses of relevant, local organizations, and networks are also included. The information material is also included in the report sent to the General Practitioner (GP) and home care.
  Interventions: Behavioral: Empowerment
- Conversation with Nurse (Other): Patients in the intervention group 2 gets clarification and follow-up conversation with a nurse anchored in both medical department and municipalities. The nurse is "blinded" in relation to the patient's screening results. Problems identified in connection therewith are communicated to the GP and home care.
  Interventions: Other: Conversation with nurse
- Controle Group (No Intervention): Patients in the control group are undergoing the same measurements and records at discharge, as the intervention group, but are otherwise receiving treatment and care as usual without further intervention.

INTERVENTIONS:
Behavioral: Empowerment — To give patients the necessary resources to take care of their own health
  Arms: Empowerment
Other: Conversation with nurse — To find out, if the nurse, using her ....
  Arms: Conversation with Nurse

SUMMARY:
Randomized Clinical Trial (RCT) To investigate and compare the effect of two preventive interventions on readmission rates, loss of functions, quality of life and cost-benefit.

DETAILED DESCRIPTION:
At baseline:

Nutritional status, BMI and weight, depression (GDS5), dementia (MMSE), pain (Verbal Ranking Scale), muscle strength (hand-grip strength, chair-to-stand-test), quality of life (EQ5D), coping (Sense of Coherence 13 item scale), patient experience (NORPEQ), medication management (MedMaide).

At follow-up three months after discharge:

BMI and weight, depression (GDS5), dementia (MMSE), pain (Verbal Ranking Scale), muscle strength (hand-grip strength, chair-to-stand-test) and EQ5D. In addition, need for initiated municipal assistance after discharge. Project employee who performs data collection is blinded to the group to which the patient is randomized.

The control group Patients in the control group undergo the same measurements and registrations at discharge and 3 - month follow-up, as the intervention groups, but receive otherwise usual treatment and care, and are discharged without further intervention. After six months control patients receive a report comprising the screening results, relevant information material and a cover letter. Patients' GP and municipality care section receive a summary of outcomes, as well as a cover letter.

Register data Information on mortality, readmissions and services in primary health care are obtained after 6 months from the National Patient Register, Population Register and municipalities.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* Living in their own home with no contact to the Municipality, both before and after admission
* Discharged from Department o105 or the Acute Receiving Unit <48 hours from admission.

Exclusion Criteria:

* Patients with life-threatening disease in the terminal stage
* Patients who does not speak and understand Danish
* Patients who are not able to communicate and collaborate, with regards to the measurements

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of participants who have been readmitted to hospital | 01.03.2013 - 12.31.2014
  Number of participants who have been readmitted to hospital. Measured 6 months after admission.

SECONDARY OUTCOMES:
Mortality | 01.04.2014 - 31.12.2014
  Mortality. Number of participants, who have died. Measured 6 months after admission.
Functional ability | 31.12.2014
  Measured 3 months after discharge.
  Functional ability
  Handgrip-strength 4 second test: Hand- and forearm muscular strength in kg. and 30 second chair stand test: Lower-body muscle strength
Primary Healthcare Services | 01.04.2013 - 31.12.2014
  Delivered services in Primary Healthcare. Measured 6 months after admission.

CONTACTS AND LOCATIONS:
Overall Officials: Tove L. Damsgaard, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark